CLINICAL TRIAL: NCT04718506
Title: Rehabilitation for Post-COVID-19 Syndrome Through a Multicomponent, Educational and Supervised Exercise Intervention [RECOVE]
Brief Title: Rehabilitation for Post-COVID-19 Syndrome Through a Supervised Exercise Intervention
Acronym: RECOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Javier Courel Ibáñez, Principal Investigator, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3036/2020
Record Dates: First submitted 2021-01-16; First posted 2021-01-22 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Covid19; Post-COVID-19 Syndrome
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise (Experimental): Supervised exercise training
  Interventions: Behavioral: Exercise
- Inspiratory muscle training (Experimental): Non-supervised inspiratory muscle training protocol
  Interventions: Behavioral: Controls
- Controls (Active Comparator): Non-supervised WHO exercise guidelines
  Interventions: Behavioral: Inspiratory muscle training

INTERVENTIONS:
Behavioral: Exercise — Participants from the experimental group will complete 8 weeks of a tailored, educational and supervised multicomponent exercise program adapted from the ACSM guidelines for Chronic Obstructive Pulmonary Disease and Cardiovascular Disease. Participants will complete a 3-days-a-week concurrent training routine: two days of resistance training (50% 1RM (one-repetition maximum), 3 sets, 8 repetitions, 4 exercises [squat, bench press, deadlift and bench pull]) combined with Moderate Intensity Variable Training (MIVT: 4-6 x 3-5 min at 70-80% Heart Rate Reserve (HRR) / 2-3 min at 55-65% HRR), and one day of Light Intensity Continuous Training (LICT: 30-60 min, 65-70% HRR). Progressions will be individualized and consistent with patient tolerance. Sessions will be supervised by certified strength and conditioning coaches, Graduated in Sports Sciences
  Arms: Exercise
Behavioral: Inspiratory muscle training — Participants enrolled in the inspiratory muscle training protocol will used the PowerBreath® Classic Heath Series mechanic threshold devices to perform 1 set of 30 repetitions, twice a day, every day of the week. This assumes a work intensity of approximately 62.5% ± 4.6% of the PIM (maximum inspiratory pressure). Increase in resistance will be made every two weeks by turning the load adjustment clockwise ¼ to 1 full turn, pending on participant tolerance to maintain a 12-15 RPE on modified Borg scale. The training will be preceded by a warm-up at 80% of the 30 RM load, with 2 min of rest between sets
  Arms: Controls
Behavioral: Controls — Controls will be advised (non-supervised) to follow the WHO guidelines: Support for Rehabilitation: Self-Management after COVID-19 Related Illness
  Arms: Inspiratory muscle training

SUMMARY:
This is a randomized controlled trial of the efficacy of a tailored exercise program, based on multicomponent exercise training and/or inspiratory muscle training, compared to the WHO self-management leaflet commonly used in outpatient scenarios, on the recovery of persistent symptoms and functional limitations after COVID-19.

. The primary objective of the study is to evaluate the clinical efficacy and safety of a tailored exercise-based treatment relative to the control arm in improving the subject clinical status in ambulatory patients.

DETAILED DESCRIPTION:
A fraction ~10% of the COVID-19 patients who undergo a variable acute symptomatic phase of the disease are coming forward with continuing effects of the disease over a month, with chronic complaints like mental fog, delayed latent periods in recalling events of recent past, tachycardia, extreme fatigue, inability to perform daily physical tasks and likely to develop stress, depression, irritability, insomnia, fear, confusion, anger and frustration. This condition is defined as post-COVID-19 syndrome and increasingly affecting a high number of people as the pandemic evolves.

The post-COVID-19 syndrome has become a usual situation in the evolutionary course of the disease with its own entity. The National Health Service (NHS) of UK has recently published a clinical guide for long-term management of the effects of COVID-19 with a comprehensive plan for the assessment and care of patients who present or develop symptoms from the fourth week after diagnosis.

The effective long-term management of the effects of COVID-19 is a challenge that requires awareness. The RECOVE project aims at determining the role of exercise in the treatment of post-COVID-19 syndrome ambulatory patients.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 diagnosed using real-time reverse transcriptase polymerase chain reaction (PCR) tests or positive for SARS-CoV-2 virus antigen >90 days before randomization.
* Still present a chronic symptomatic phase lasting >90 days since debut of symptoms
* Have not been hospitalized
* There is no evidence on clinical records of pneumonia or any other organ failure related to SARS-CoV-2
* Non-coincident participation in any intervention trial
* Capable and willing to provide an informed consent

Exclusion Criteria:

* Refusal to participate expressed by patient or legally authorized representative if they are present
* Pregnancy or breast-feeding.
* Acute heart attack (recent 3-6 months) or unstable angina
* Uncontrolled atrial or ventricular arrhythmias
* Aortic dissecting aneurysm
* Severe aortic stenosis
* Acute endocarditis / pericarditis
* Uncontrolled high blood pressure (>180/100 mmHg)
* Acute thromboembolism
* Acute or severe heart failure
* Acute or severe respiratory failure
* Uncontrolled acute decompensated diabetes mellitus or low blood sugar
* A recent fracture in the last month.
* Conditions preventing cooperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2022-02-06 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Changes in subject clinical status | Baseline to 8 Weeks
  Post-COVID Functional Status (PCFS) on a 5-point ordinal scale (0 to 4 grades) and medical screening

SECONDARY OUTCOMES:
Changes in cardiovascular fitness: Maximal oxygen consumption (VO2max) | Baseline to 8 Weeks
  VO2max estimated from standard algorithms using a submaximal multistage and individualized cardiopulmonary exercise test on cycloergometer. Heart rate (HR), rate of perceive effort (RPE) and load (W) will be combined to report VO2max in mml/kg/min.
Changes in neuromuscular performance during resistance exercise: Barbell Mean Propulsive Velocity (MPV) | Baseline to 8 Weeks
  Barbell displacement and velocity will be monitored in real time using a linear transductor during a progressive resistance training exercise tests. Displacement and velocity will be combined to report MPV
Changes in balance: center of pressure (COP) sway | Baseline to 8 Weeks
  COP sway during a balance test will be measured using a high resolution force plate
Changes in pulmonary function: Forced Vital Capacity (FVC) | Baseline to 8 Weeks
  The total amount of air exhaled (mL) during a forced expiratory volume test will be measured by spirometry.
Changes in pulmonary function: Forced expiratory volume (FEV) | Baseline to 8 Weeks
  The amount of air exhaled (mL) during the first (FEV1), second (FEV2), and third seconds (FEV3) of the forced breath will be measured by spirometry.
Changes in high sensitivity C-reactive protein (hsCPR) | Baseline to 8 Weeks
  hsCPR (mg/L) determined by blood-based biochemistry analysis
Changes in D-dimer | Baseline to 8 Weeks
  D-dimer (mg/L) determined by blood-based biochemistry analysis
Changes in Troponin | Baseline to 8 Weeks
  Troponin (ng/mL) determined by blood-based biochemistry analysis
Changes in glutamic-pyruvic transaminase (GPT) | Baseline to 8 Weeks
  GPT(IU/L) determined by blood-based biochemistry analysis
Changes in serum creatine kinase (CK) | Baseline to 8 Weeks
  CK (U/L) determined by blood-based biochemistry analysis lactate dehydrogenase (LDH)
Changes in lactate dehydrogenase (LDH) | Baseline to 8 Weeks
  LDH (U/L) determined by blood-based biochemistry analysis
Changes in physical activity levels | Baseline to 8 Weeks
  Metabolic Equivalents (METs) throughout a week, including activity for work, during transport and leisure time, using the self-reported general physical activity questionnaire (GPAQ)
Changes in tolerance to exercise: DePaul Symptom Questionnaire for Post-exertional malaise (DSQ-PEM) scores | Baseline to 8 Weeks
  DSQ-PEM will be administrate to obtain a score of tolerance to exercise (DSQ-PEM Scoring depends on the 10-item mixed questionnaire including scale and yes/no questions)
Changes in fatigue: Chalder Fatigue Scale scale (CFQ-11) | Baseline to 8 Weeks
  CFQ-11 will be administrate to obtain a score of fatigue (Each of the 11 items are answered on a 4-point scale ranging from the asymptomatic to maximum symptomology)
Changes in anxiety: Generalized Anxiety Disorder scale (GAD7) | Baseline to 8 Weeks
  GAD7 will be administrate to obtain a score of anxiety status (total score for the seven items ranges from 0 to 21)
Changes in depression: Patient Health Questionnaire (PHQ9) | Baseline to 8 Weeks
  PHQ9 will be administrate to obtain a score of depression status (total score for the nine items ranges from 0 to 27)
Changes in health related quality of life: 12-item Short Form Survey (SF12) | Baseline to 8 Weeks
  Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). The scores will be reported as Z-scores (difference compared to the population average, measured in standard deviations).

OTHER OUTCOMES:
Changes in Percent Body Fat | Baseline to 8 Weeks
  Body composition will be measured by bioelectrical impedance analysis

CONTACTS AND LOCATIONS:
Overall Officials: Javier Courel-Ibáñez, Ph.D, Principal Investigator — Faculty of Sport Sciences, University of Murcia, Spain.; Amaya Jimeno-Almazán, Dr,, Principal Investigator — University Hospital of Santa Lucía, Infectious Diseases Section,; Jesús García Pallarés, Ph.D, Study Director — Faculty of Sport Sciences, University of Murcia, Spain.
Locations (1):
- Faculty of Sport Sciences, Murcia, San Javier, Spain